CLINICAL TRIAL: NCT01317966
Title: A Multicentre Investigation of Recombinant Human Interleukin-11 (rhIL-11) Combination Low-dose Rituximab in Management of Steroid-Resistant/Relapsed Immune Thrombocytopenia (ITP)
Brief Title: Recombinant Human Interleukin-11 Combination Low-dose Rituximab in Immune Thrombocytopenia
Acronym: Incritop
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patients were enrolled.
Sponsor: Ming Hou (Other)
Collaborators: Peking Union Medical College Hospital (Other); Chinese Academy of Medical Sciences (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); West China Hospital (Other); Shandong Provincial Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Ming Hou, Director of Hematology Department, Shandong University
Organization: Shandong University (Other)
Other Study IDs: ITP-001
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2011-11

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — oprelvekin; Rituximab; Inosine Triphosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rhIL-11Combinating Low-dose Rituximab: rhIL-11 (interleukin-11, Juheli) 50 mcg/kg subcutaneously daily for 14 days
  Rituximab 100mcg weekly for 4 weeks
  Interventions: Drug: rhIL-11

INTERVENTIONS:
Drug: rhIL-11 — Recombinant Human Interleukin-11 (rhIL-11) Combinating Low-dose Rituximab
  Other Names: Rituximab; ITP

SUMMARY:
The purpose of this study is to determine whether Recombinant Human Interleukin-11 (rhIL-11) Combination Low-dose Rituximab prednisone are effective and safe in the management of Steroid-Resistant/Relapsed Immune Thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

1. Patients may be male or female, between the ages of 16 ~ 75 years old.
2. Isolated thrombocytopenia with an otherwise normal peripheral blood smear and no other causes of thrombocytopenia, morphologically normal bone marrow aspirate with normal to increased number of megakaryocytes, and absence of splenomegaly.
3. To show a platelet count ≤ 30 × 109/L, or platelet count ≥ 30 × 109/L with bleeding manifestations at the moment of the first infusion with the study product.
4. ＥＣＯＧ performance status ≤ 2.
5. Patients failed to respond to acceptable dose of steroids for 4 weeks, or relapsed. Some patients were also refractory to splenectomy.
6. Patients must be willing and able to give written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia).
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator (or coinvestigator).

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response (Complete Response) | The time frame is up to 14 days per subject
  CR. A complete response (CR) was defined as a sustained (≥ 4 months) platelet count ≥ 100×109/L without recurrence of thrombocytopenia

SECONDARY OUTCOMES:
Evaluation of platelet response (R) | The time frame is up to 14 days per subject
  R. A response (R) was defined as a sustained (≥ 4 months) platelet count ≥ 30×109/L without recurrence of thrombocytopenia
The time of rhIL-11 onset. | The time frame is up to 28 days per subject.
  The time to platelet recovery (deﬁned as the number of days from the start of the study to the ﬁrst day with a platelet count of ≥30 × 109/L)
DFS | The time frame is up to 90 days per subject.
  The median disease-free survival periods
The number and frequency of IL-11 associated adverse events. | up to 14 days per subject

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Result] Zaja F, Vianelli N, Volpetti S, Battista ML, Defina M, Palmieri S, Bocchia M, Medeot M, De Luca S, Ferrara F, Isola M, Baccarani M, Fanin R. Low-dose rituximab in adult patients with primary immune thrombocytopenia. Eur J Haematol. 2010 Oct;85(4):329-34. doi: 10.1111/j.1600-0609.2010.01486.x. Epub 2010 Jul 28. PMID 20546023